CLINICAL TRIAL: NCT06847633
Title: A Digital Lifestyle Intervention in Primary Healthcare to Prevent Cardiovascular Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Capio Narsjukvard (Unknown)
Responsible Party: Principal Investigator, Marie Löf, docent, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-07911-01
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Diseases; Lifestyle Factors
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital lifestyle intervention (Experimental): Access to the digital intervention which will provide support for healthier lifestyle behaviors regarding diet, physical activity, sleep, stress, alcohol consumption, and use of tobacco.
  Interventions: Behavioral: Digital lifestyle intervention
- Control arm (No Intervention): Standard care i.e., a routine appointment to the primary healthcare center for discussing lifestyle habits

INTERVENTIONS:
Behavioral: Digital lifestyle intervention — The digital lifestyle intervention provides support to the patient through digital lectures, home assignments and digital group meetings as well as provides the possibility for the healthcare provider to provide personalized digital support and feedback to the patient
  Arms: Digital lifestyle intervention

SUMMARY:
Unhealthy lifestyle behaviors are well-established risk factors for cardiovascular disease (CVD) which is the leading cause of death globally and in Sweden. Digitalization offers new and better possibilities for healthcare to fulfil their responsibility to support healthier lifestyles, however, to ensure scalability and sustained implementation of digital tools within healthcare, digital interventions need to be systematically maintained and delivered by the primary healthcare. The aim of this project is to evaluate whether a digital lifestyle intervention, developed within Swedish primary healthcare, can improve clinically important cardiovascular health outcomes and lifestyle behaviors. In this multi-center randomized controlled trial patients, 40-60 years, in Swedish primary healthcare will be recruited and randomized to the control or intervention group. All participants will receive standard care consisting of one structured health dialogue focused on lifestyle habits. The intervention group will also receive support through the digital lifestyle intervention for creating healthy habits regarding diet, physical activity, alcohol consumption, and tobacco usage. The primary outcome is LDL-cholesterol at 6 months post-randomization. Secondary outcomes 6 months post-randomization are HDL-, total cholesterol, fasting blood glucose, triglycerides, non-HDL, blood pressure, weight, height, BMI, waist circumference, cardiovascular risk evaluation (SCORE2), dietary intake, physical activity, sleep, stress, alcohol consumption, tobacco use, and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Attended a Health dialogue visit to primary healthcare for patients 40-60 years old
* Willing to change at least one lifestyle behavior regarding physical activity, diet, smoking/snus, alcohol, sleep, or stress

Exclusion Criteria:

* diabetes
* heart failure
* history of myocardial infarction
* history of stroke
* pregnancy

Ages: 39 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
LDL-cholesterol | 6 months post-randomization
  Low density lipoprotein cholesterol

SECONDARY OUTCOMES:
HDL-cholesterol | 6 months post-randomization
  High density lipoprotein cholesterol
Total cholesterol | 6 months post-randomization
Fasting blood glucose | 6 months post-randomization
Triglycerides | 6 months post-randomization
Non-HDL cholesterol | 6 months post-randomization
  Calculated by subtracting HDL cholesterol from total cholesterol
Systolic blood pressure | 6 months post-randomization
Diastolic blood pressure | 6 months post-randomization
Weight | 6 months post-randomization
Height | 6 months post-randomization
Body mass index | 6 months post-randomization
Waist circumference | 6 months post-randomization
Systematic COronary Risk Evaluation model, second version (SCORE2) | 6 months post-randomization
  Estimated percentage risk of fatal and non-fatal cardiovascular disease within the next 10 years. The estimation is based on data on sex, age, smoking, systolic blood pressure (SBP), total cholesterol, and HDL cholesterol
Health-related quality of life | 6 months post-randomization
  Measured by the questionnaire EuroQol-5 Dimensions-5 Levels (EQ-5D-5L). Five dimensions including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five response options, scored 1-5, ranging from 'no problems' to 'extreme problems'
Health-related quality of life | 6 months post-randomization
  Measured by the questionnaire EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) visual analogue scale (VAS) ranging from 0 to 100 where higher values represents better self-assessed health.
Diet intake | 6 months post-randomization
  Assessed by questions on intake quantity of vegetables, fruit, sweet beverages, and snacks the past week
Physical activity | 6 months post-randomization
  Assessed by questions on time (minutes and hours) spent in moderate and vigorous physical activity the past week
Sedentary time | 6 months post-randomization
  One question about time in sitting position
Stress | 6 months post-randomization
  Assessed by the Perceived Stress Scale. Minimum value 0. Maximum value 56. Higher scores indicating greater perceived stress.
Sleep | 6 months post-randomization
  Assessed by the Karolinska Sleep Questionnaire. No single set of minimum and maximum values. Each item is scored from 0-5, where higher values indicate greater sleep issues
Alcohol consumption | 6 months post-randomization
  Questions on monthly frequency of heavy episodic drinking, weekly alcohol consumption
Tobacco use | 6 months post-randomization
  Questions on frequency of smoking and using snus the past week and the past 4 weeks
Mediated effects on behavior change | 6 months post-randomization
  Potential mediators to be assessed are confidence, importance, and know-how (i.e., knowing how to change a behavior).
Participant experience from using the digital intervention | 6 months post-randomization
  Questions on experience from using the intervention (intervention group only). The questions are framed as statements with five response options ranging from 'Not agreeing at all' to 'Fully agreeing'

CONTACTS AND LOCATIONS:
Overall Officials: Marie Löf, PhD, Principal Investigator — Karolinska Institutet
Locations (6):
- Sweden (6):
  - Primary helathcare centers in Region Gävleborg, Gävle
  - Primary healthcare centers in Region Halland, Halmstad
  - Primay healthcare centers in Region Östergötland, Linköping
  - Primary healthcare centers in region Skåne, Malmo
  - Primary healthcare centers in Region Västerbotten, Umeå
  - Primary healthcare centers in Region Västmanland, Västerås

IPD SHARING:
Plan to Share IPD: No